CLINICAL TRIAL: NCT04292457
Title: Namsos Anaesthesia Children Outcome Study (NACOS)
Brief Title: Namsos Anaesthesia Children Outcome Study
Acronym: NACOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: ØNH Legen Trondheim (Unknown); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43654
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Emergence Delirium
Keywords: Pediatric Anaesthesia; Emergence Delirium; Postoperative Behavioral Changes; Sevoflurane; Propofol; Adenotonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Experimental): Anesthesia is maintained with Propofol
  Interventions: Drug: Propofol
- Sevoflurane (Experimental): Anesthesia is maintained with Sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Anesthesia is maintained with a continuous infusion of Propofol. Induction of anesthesia and anesthetic management are otherwise the same in both study arms.
  Arms: Propofol
Drug: Sevoflurane — Anesthesia is maintained with a continuous inhalation of Sevoflurane. Induction of anesthesia and anesthetic management are otherwise the same in both study arms.
  Arms: Sevoflurane

SUMMARY:
Behavioral disturbances are often seen in children after anesthesia both immediately after surgery (emergence delirium) and after discharge from hospital. Persisting behavioral changes may affect emotional and cognitive development. It is known that both type of surgery and anesthetic management affect the occurrence of behavioral disturbances. Specifically, differences in occurrence were found after sevoflurane anesthesia and propofol anesthesia, two anesthetics that are generally used in practice. However, evidence is based on methodologically weak studies.

The described occurrence of behavioral disturbances in children after anesthesia is not in line with the investigators' clinical experience, and neither are the described differences in occurrence between sevoflurane anesthesia and propofol anesthesia. This study will compare emergence delirium and behavioral changes after discharge from hospital in children who had surgery for removal of their tonsils under sevoflurane anesthesia versus propofol anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* adenotomy and/or tonsillotomy and/or tonsillectomy
* ASA physical status class I or II

Exclusion Criteria:

* unexperienced ear-nose-throat (ENT) surgeon (ENT surgeon < 1 year of training, ENT surgeon without experience with the use of laryngeal mask as airway during adenotomy/tonsillotomy/tonsillectomy)
* preoperative syndromes
* ASA physical status class > 2
* missing written consent from parents/guardians

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 761 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium Scale (PAED) ≥ 10 | 1 hour
  A PAED score ≥ 10 during the first hour after emergence from anaesthesia is defined as an ED event occuring

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability Scale (FLACC) ≥ 4 | 1 hour
  A FLACC score ≥ 4 during the first hour after emergence from anaesthesia is defined as moderate or severe pain
Post Hospital Behavioral Questionnaire (PHBQ) | 7 days
  An average score > 3 in one or more of the questionnaire categories is defined as postoperative behavioural change
Post Hospital Behavioral Questionnaire (PHBQ) | 30 days
  An average score > 3 in one or more of the questionnaire categories is defined as postoperative behavioural change

CONTACTS AND LOCATIONS:
Overall Officials: Hallvard Græslie, MD, Study Chair — Head of surgical Clinic, Namsos Hospital, Nord-Trondelag Hospital Trust
Locations (2):
- Norway (2):
  - Namsos Hospital, Nord-Trondelag Hospital Trust, Namsos, Trøndelag
  - ØNH Legen, Trondheim, Trøndelag

IPD SHARING:
Plan to Share IPD: Undecided